CLINICAL TRIAL: NCT07042945
Title: Multiple Dose Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiretroviral Activity of MK-4646 Monotherapy in Antiretroviral Therapy-Naïve Participants With HIV-1
Brief Title: MK-4646 Multiple Dose Trial in Participants With Human Immunodeficiency Virus Type 1 (HIV-1) (MK-4646-003)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4646-003; MK-4646-003 (Other: MSD); 2025-521102-17-00 (Registry Identifier: EU CT); U1111-1318-7985 (Registry Identifier: UTN)
Record Dates: First submitted 2025-06-09; First posted 2025-06-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- MK-4646 Panel A (Experimental): MK-4646 160 mg every 24 hours (q24h) for 7 days
  Interventions: Drug: MK-4646
- MK-4646 Panel B (Experimental): MK-4646 ≤460 mg q24h for 7 days
  Interventions: Drug: MK-4646
- MK-4646 Panel C (Experimental): MK-4646 ≤460 mg q24h for 7 days
  Interventions: Drug: MK-4646
- MK-4646 Panel D (Experimental): MK-4646 ≤460 mg every 12 hours (q12h) for 7 days
  Interventions: Drug: MK-4646

INTERVENTIONS:
Drug: MK-4646 — MK-4646 in capsular form administered orally

SUMMARY:
This study will examine if at least one dose level of MK-4646 can lower HIV-1 viral load in a person's blood by a certain amount. The goals of this study are to learn about the safety of MK-4646 and if people tolerate it; and how HIV-1 viral load may decrease after starting to take MK-4646.

ELIGIBILITY:
Inclusion Criteria:

* Other than having HIV-1, is in good health
* Is antiretroviral therapy (ART)-naïve
* If ART-experienced has not received any antiretroviral therapy within 60 days (or 5 half-lives, whichever is longer) prior to screening
* Is willing to receive no other ART prior to Day 8 post-dose of the trial
* If capable of producing sperm agrees to use contraception
* If assigned female sex at birth is not breastfeeding
* A participant of childbearing potential (POCBP) is not pregnant and has a negative highly sensitive pregnancy test (urine or serum), and uses a contraceptive method that is highly effective

Exclusion Criteria:

* Has acute (primary) HIV-1 infection
* Has history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years.
* Has history of cancer (malignancy)
* Has history of significant multiple and/or severe allergies
* Tests positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies
* Has had a major surgery and/or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit
* Has received any vaccine starting from 30 days prior to study intervention or is scheduled to receive any vaccine through 14 days following study intervention
* Is unable to refrain from using protocol specified prohibited medications
* Is an excessive smoker, or consumes excessive amounts of alcoholic or caffeinated beverages
* Is a regular user of any illicit drugs or has a history of drug (including alcohol) abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Participants with averse events (AEs) | 14 days post last dose (Up to Day 23)
  Percentage of participants with one or more AEs
Participants who discontinued study medication due to an AE | Up to Day 7
  Percentage of participants who discontinued study medication due to an AE
Viral load decline of plasma HIV-1 ribonucleic acid (RNA) | Predose, 1,2, 3, 4 and 5 days postdose
  Time course of plasma HIV-1 RNA viral load decline.

SECONDARY OUTCOMES:
Area under the curve from time 0 to 24 hours (AUC0-24) of MK-4646 | Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose
  AUC0-24 postdose of plasma MK- 4646 in the fasted state
Maximum plasma concentration (Cmax) of MK-4646 | Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose
  Cmax postdose of plasma MK- 4646 in the fasted state
Concentration at 24 hours (C24) of MK-4646 | 24 hours postdose
  C24 postdose of plasma MK- 4646 in the fasted state
Time to maximum concentration (Tmax) of MK-4646 | Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose
  Tmax postdose of plasma MK- 4646 in the fasted state
Half life (t1/2) of MK-4646 | Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24 hours postdose
  T1/2 postdose of plasma MK- 4646 in the fasted state

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- PMSI Republican Clinical Hospital "T.Mosneaga" ( Site 0002), Chisinau, Moldova
- ARENSIA Exploratory Medicine ( Site 0001), Bucharest, București, Romania

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com